CLINICAL TRIAL: NCT00468260
Title: An Open Label Phase I Study to Evaluate the Effects of Patupilone on the Pharmacokinetics and Pharmacodynamics of Warfarin in Patients With Advanced Malignancies-extension Study
Brief Title: The Effects of Patupilone on the Pharmacokinetics and Pharmacodynamics of Warfarin in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: pts. will be captured in core
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2120E1
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Advanced Malignancies
Keywords: Cancer; EPO906; Patupilone
MeSH Terms: conditions — Neoplasms | interventions — epothilone B

INTERVENTIONS:
Drug: Patupilone

SUMMARY:
To evaluate the effects of patupilone on the pharmacokinetics of warfarin in patients with advanced malignancies.

ELIGIBILITY:
Inclusion criteria Participation in study EPO906A2120E1

* Age ≥ 18 years of age
* Life expectancy ≥ 3 months
* Histologically documented advanced solid tumors which have progressed after standard systemic therapy or for which standard systemic therapy does not exist
* Completed all PK sampling in the core study

Exclusion criteria

* Known diagnosis of human immunodeficiency virus (HIV) infection, hepatitis
* Female patients who are pregnant or breast feeding
* Patients with a severe and/or uncontrolled medical disease

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-05

PRIMARY OUTCOMES:
Safety
Tolerability
Potential activity of patupilone once every 21 days in patients that completed the core study

SECONDARY OUTCOMES:
Objective response and tumor evaluation assessed by response evaluation criteria in solid tumors (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- San Antonio, Texas, United States